CLINICAL TRIAL: NCT00857870
Title: Comparative Investigation of Efficacy and Safety of Insulin Glargine Versus Metformin as First Line Drug in Treatment of Early Type 2 Diabetes
Brief Title: Insulin Glargine First Line vs Metformin in Type 2 Diabetic Subjects
Acronym: GLORY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GWT-TUD GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GWT-2008-1
Record Dates: First submitted 2009-03-06; First posted 2009-03-09 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Insulin Glargine

ARMS (2):
- Metformin (Active Comparator)
  Interventions: Drug: Metformin
- Insulin glargine (Active Comparator)
  Interventions: Drug: Insulin glargine

INTERVENTIONS:
Drug: Metformin — Metformin is administered as coated tablet. Initial dose is 500 mg twice a day (morning and evening) during or after the meal. The first administration takes place on the evening of visit 1c. The duration of the therapy is 36 weeks until visit 8c.
  Initial dose of 500 mg bid was increased after 4 weeks (visit 2) to 850 mg bid when the patient tolerated the initial dose. If the side effects were not tolerable, the initial dose was decreased to 500 mg once a day and where appropriate increased at a later visit.
  After 8 weeks (visit 3) metformin dose was increased to 1000 mg bid when tolerated. If dose is not tolerated, it was decreased to the next lower dose.
  Arms: Metformin
Drug: Insulin glargine — Insulin glargine is given subcutaneously with an insulin-pen (SoloStar®). The dose was titrated to reach a fasting plasma glucose value of <5.6 mmol/l. Insulin glargine was given once a day in the evening before going to bed (bed-time injection). The first insulin injection takes place on the evening of visit 1c. The duration of the therapy is 36 weeks until visit 8c. All patients were trained in handling and storage of the insulin-pen.
  Arms: Insulin glargine

SUMMARY:
Comparison of efficacy and safety of glargine insulin and metformin as first line drug of patients insufficiently treated with lifestyle intervention. So far treatment also algorithm with lifestyle and metformin has not been evaluated in patients with type 2 diabetes and HbA1C greater or equal 7 % and lower than 8.1%.Besides HbA1C postprandial glucose excursion and glycemic variability as determinants of oxidative stress will be measured by continuous glucose measurement(CGM). Further more CGM will reveal risk of hypoglycemia at night. As secondary objectives effect on endothelial function, renal function and biomarkers of low great inflammation will be evaluated. So far only scarce information on face to face comparison in ealy diabetes exists.

ELIGIBILITY:
Inclusion Criteria:

* early type 2 diabetes (lower than 5 years known)
* male and female(35 to 75 years)
* HbA1c 7 to 8 %, if drug naive and <= 8.5 with previous OAD intake
* Informed consent

Exclusion Criteria:

* any treatment more than one OAD at the same time
* treatment with one OAD < 6 weeks time
* insulin treatment
* acute coronary syndrome < 6 months
* severe liver disease
* alcohol abuse or drug addiction
* severe kidney disease
* acute critical illness with renal impairment
* i.v. application of iodine
* ketoacidosis
* acute or chronic illness witch may lead to hypoxia or cardial failure
* allergy against one of the drugs
* deficit in compliance or cooperation
* pregnancy or breast feeding
* women in fertile age without accepted contraceptive

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2009-03; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) after a testmeal measured CGM. | baseline and visit 8

SECONDARY OUTCOMES:
HbA1C, glycemic variability, glycemic load, insulin secretion after testmeal, free fatty acids, biomarkers of low grade inflammation, endothelial dysfunction. | baseline and visit 8

CONTACTS AND LOCATIONS:
Locations (1):
- GWT -TUD, Center for Clinical Studies, Dresden, Germany

REFERENCES:
- [Derived] Pistrosch F, Kohler C, Schaper F, Landgraf W, Forst T, Hanefeld M. Effects of insulin glargine versus metformin on glycemic variability, microvascular and beta-cell function in early type 2 diabetes. Acta Diabetol. 2013 Aug;50(4):587-95. doi: 10.1007/s00592-012-0451-9. Epub 2013 Feb 21. PMID 23430192